CLINICAL TRIAL: NCT06879678
Title: Evaluating a Web-Based Exercise Program for Neuropathic Symptoms and Quality of Life in Breast Cancer Patients Undergoing Chemotherapy: A Randomized Controlled Tria
Brief Title: Web-Based Exercise for Neuropathy and Quality of Life in Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Sabahat Coşkun, Associate Professor Dr., Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Bilecik14
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy (CIPN); Breast Cancer
Keywords: Breast Cancer; Chemotherapy-Induced Peripheral Neuropathy (CIPN); Exercise Therapy; Quality of Life; Web-Based Intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study population will consist of breast cancer patients who receive taxane-based chemotherapy and meet the inclusion criteria at the Day Chemotherapy Unit of a training and research hospital. A sample size calculation has been conducted for the study. Before conducting the power analysis, the effect size must be determined. In this study, the effect size has been derived from a similar previous study. Based on this study, the Type-1 error (α) is set at 0.05, power (1-β) is 0.85, and the effect size (d = 0.60) for the Student's t-test has been calculated. Based on these parameters, the minimum required sample size is expected to be 41 patients per group, totaling 82 participants. However, considering potential dropouts during the study, it is planned to include a total of 90 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): standard protocol
- Intervention group (Experimental): Web-Based Exercise Program + standard protocol
  Interventions: Behavioral: Web-Based Exercise Program

INTERVENTIONS:
Behavioral: Web-Based Exercise Program — Web-Based Exercise Program + standard protocol
  Arms: Intervention group

SUMMARY:
Chemotherapy is a widely used treatment method for cancer patients. However, various side effects may occur depending on the drug used, treatment duration, and dosage. One of these side effects is chemotherapy-induced peripheral neuropathy (CIPN). CIPN is a common complication that negatively affects patients' quality of life due to nerve damage.

In particular, taxane-based chemotherapy drugs (e.g., docetaxel and paclitaxel), which are commonly used in the treatment of breast cancer, can lead to peripheral neuropathy. Studies indicate that the incidence of taxane-induced neuropathy ranges between 61% and 92%. While this condition primarily presents with sensory symptoms, it can also affect motor and autonomic nervous system functions in some patients.

Currently, pharmacological treatments for preventing CIPN are limited. Aside from duloxetine, no medication has been proven effective. Therefore, non-pharmacological approaches, such as exercise, are considered an important alternative for alleviating neuropathy symptoms.

Exercise is emerging as an effective method for preventing and managing peripheral neuropathy during cancer treatment. Research suggests that regular exercise has positive effects on the nervous system and can help reduce neuropathic symptoms, thereby improving patients' quality of life.

This randomized controlled trial aims to evaluate the effects of a web-based exercise program on neuropathic symptoms and quality of life in breast cancer patients undergoing chemotherapy. The study consists of two phases: In the first phase, a web-based exercise program will be developed under the guidance of a physiotherapist to help manage neuropathic symptoms. In the second phase, the effectiveness of this program will be assessed. Data will be collected using the Patient Information Form, Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT), and the EORTC QLQ-C30 Quality of Life Questionnaire. Evaluations will be conducted before the intervention and at the end of an 8-week period in both the intervention and control groups.

This study aims to demonstrate the potential effects of web-based exercise programs in alleviating neuropathic symptoms and improving quality of life in cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer among women worldwide and in our country, ranking second among the leading causes of cancer-related deaths. Chemotherapy drugs are among the most widely used treatment methods for breast cancer. Peripheral neuropathy (PN) is one of the most common side effects caused by chemotherapy drugs, characterized by damage to the nervous system. This condition is specific to all chemotherapy drug classes and can develop even after a single drug administration. However, in most cases, it increases depending on the dose and duration of the drug, especially in elderly patients, those with diabetes, alcohol users, individuals with metabolic disorders, and those with vitamin B12 deficiency. Furthermore, the mechanisms responsible for the development of peripheral neuropathy have not yet been thoroughly elucidated.

The clinical symptoms of chemotherapy-induced peripheral neuropathy (CIPN) include tingling, numbness, muscle weakness, loss of balance, changes in touch, pain, and temperature perception, as well as constipation, postural hypotension, and loss of deep tendon reflexes. The early detection of CIPN symptoms can prevent disability, falls, and injuries, minimizing the progression of symptoms and complications. Otherwise, the presence and severity of neuropathic pain can negatively impact walking, daily activities, sleep, work, mood, enjoyment of life, and interpersonal relationships. This, in turn, can lead to a decline in patients' quality of life. Additionally, in patients experiencing these issues, dose reductions, treatment cancellations, or delays can adversely affect the treatment process and survival rates. In this context, the inability to tolerate the full dose and duration of chemotherapy due to CIPN emerges as a significant oncological issue.

There is limited evidence-based intervention to continue treatment and prevent or alleviate CIPN. Therefore, more research is needed on non-pharmacological supportive strategies to manage the burden of CIPN and improve patients' quality of life. One of the interventions with the potential to prevent or alleviate CIPN and consequently improve quality of life is exercise rehabilitation. Exercise programs play an important role in managing chemotherapy-induced side effects and improving patients' physical fitness and quality of life. Moreover, exercise programs have been found to positively impact peripheral nerves, inducing beneficial changes in vascular and metabolic systems, stimulating blood flow, and contributing to oxygen delivery.

Additionally, women who engage in moderate to vigorous physical activity before chemotherapy treatment have a lower risk of developing CIPN. Evidence-based studies have tested the positive effects of different types of exercise (aerobic, endurance, balance, and motor-sensory exercises) in reducing CIPN symptoms and improving quality of life. Most cancer patients receive chemotherapy on an outpatient basis and must manage the side effects that develop after treatment at home. During this process, cancer patients often lack professional support. Therefore, cancer patients and their families need to be supported not only in hospital settings but also at home.

Recently, there has been a rapid increase in the number of web-based education programs developed for cancer patients, which have been shown to be effective in increasing patients' knowledge levels, providing psychosocial support, reducing anxiety and depression levels, and improving quality of life. A randomized controlled web-based and mobile-supported intervention developed for women with breast cancer has been found beneficial in managing symptoms related to chronic pain and lymphedema. Furthermore, it has been observed that breast cancer patients can easily use web-based education programs and find them informative for both themselves and their families.

In this context, web-based educational programs and applications can provide interactive, cost-effective, efficient, and appropriate content for all users, including patients, families, and healthcare professionals. Delivering exercise training and follow-ups via the web can be a significant advantage for patients facing transportation difficulties, those with various physical barriers, or those who prefer the comfort and convenience of home. Planning web-based programs according to the needs of cancer patients can enhance their usage rates and effectiveness.

This study has been designed as a randomized controlled trial to evaluate the effectiveness of a web-based exercise program on neuropathic symptoms and quality of life in breast cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and speak Turkish,
* Over 18 years of age,
* Receiving taxane-based chemotherapy in daytime chemotherapy units,
* Reporting at least one neuropathy symptom according to CIPNAT,
* Diagnosed with stage II-III breast cancer,
* Receiving a planned weekly taxane-based chemotherapy infusion dose (70-99 mg/m², 100-129 mg/m², 130-159 mg/m², 160 mg/m² and above) and completing 8 treatment cycles,
* Having internet access,
* No history of deep vein thrombosis,
* Not using anticoagulant medication,
* Willing to participate in the study.

Exclusion Criteria:

* Younger than 18 years or older than 75 years,
* Having central nervous system disorders affecting movement, balance, sensation, or coordination,
* Presence of any skin infection, scar tissue, inflammation, or incision on the hands or ankles,
* Diagnosed with a proven cardiac condition or using medication for cardiac issues,
* Pregnant women or those in the postpartum period,
* History of polyneuropathy before chemotherapy,
* Cognitive impairment,
* Presence of metal implants in the exposure area,
* History of any other malignancy,
* Undergoing mastectomy.

Withdrawal Criteria

* Patients meeting the following conditions will be withdrawn from the study:
* Patients whose taxane treatment protocol is changed,
* Patients who wish to withdraw from the study,
* Patients with a pulse rate above 100 bpm,
* Patients receiving fewer than four weekly chemotherapy applications,
* Women without internet access or those who do not visit the website at least five times for four hours throughout the follow-up period.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) | At baseline (first visit) and at 8 weeks
  The Turkish validity and reliability of the scale were tested in breast cancer patients receiving taxane chemotherapy (n=430). The first section assesses sensory and motor symptoms (numbness, itching, burning, discomfort, cold sensitivity, pain, weakness, balance problems), with responses scored from 0 to 10. Higher scores indicate greater discomfort. In the second section, difficulties in daily activities (e.g., dressing, walking, working, exercising) are also rated from 0 to 10. The scale's overall Cronbach alpha is 0.87, with test-retest reliability ranging from 0.90 to 0.96. These results confirm that the scale is valid and reliable for the Turkish population.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | At baseline (first visit) and at 8 weeks
  The scale was adapted into Turkish in 2008, and its validity and reliability were determined in cancer patients. The scale consists of 30 items. It includes three subscales: functional, symptom, and global health status. The functional subscale includes physical function, role function, emotional function, cognitive function, and social function. The symptom subscale includes fatigue, nausea-vomiting, pain, shortness of breath, insomnia, appetite loss, constipation, diarrhea, and financial difficulties. The first 28 items of the scale are based on a 4-point Likert scale. The items are rated as follows: Never: 1- Very much: 4. Higher scores in this section indicate a higher level of functional ability or symptom severity. A lower average score on the symptom subscale indicates higher quality of life.The global health status of the scale is assessed with items 29 and 30, rated on a scale 1: very poor, 7: excellent. Higher scores in this section indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: SABAHAT COŞKUN, Doç.Dr., Study Director — Bilecik Şeyh Edebali Üniversity
Locations (1):
- Gulhane Education and Research Hospital, Ankara, 06010, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request, in accordance with ethical guidelines and with participant consent.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Odynets T, Briskin Y, Todorova V. Effects of Different Exercise Interventions on Quality of Life in Breast Cancer Patients: A Randomized Controlled Trial. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419880598. doi: 10.1177/1534735419880598. PMID 31625419
- [Background] Comez S, Karayurt O. The effect of web-based training on life quality and spousal adjustment for women with breast cancer and their spouses. Eur J Oncol Nurs. 2020 Aug;47:101758. doi: 10.1016/j.ejon.2020.101758. Epub 2020 Apr 9. PMID 32659714
- [Background] Bektas H, Coskun HS, Arikan F, Ozcan K, Tekeli A, Kondak Y, Sezgin MG, Yangec E, Kalav S. Development and evaluation of the efficacy of a web-based education program among cancer patients undergoing treatment with systemic chemotherapy: a randomized controlled trial. Support Care Cancer. 2022 Jul;30(7):6021-6033. doi: 10.1007/s00520-022-07039-w. Epub 2022 Apr 12. PMID 35412076
- [Background] Dixit S, Tapia V, Sepulveda C, Olate D, Berrios-Contreras L, Lorca LA, Alqahtani AS, Ribeiro IL. Effectiveness of a Therapeutic Exercise Program to Improve the Symptoms of Peripheral Neuropathy during Chemotherapy: Systematic Review of Randomized Clinical Trials. Life (Basel). 2023 Jan 18;13(2):262. doi: 10.3390/life13020262. PMID 36836620